CLINICAL TRIAL: NCT00954018
Title: Respiratory Microbial Community Composition and Metabolism in Cystic Fibrosis
Brief Title: Microbial Community Composition and Metabolism in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Thomas Martin, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 09-04-018
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — throat swabs or sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cystic Fibrosis patient during outpatient clinic visit
- Cystic Fibrosis patients during hospitalization
- CF patients about to have sinus surgery and bronchoscopy

SUMMARY:
Scientist have begun to realize that many types of bacteria often live together as a complex community, and the investigators wish to apply that idea to the bacteria in the respiratory system of people with Cystic Fibrosis (CF). It is possible that the survival of the many millions of bacteria in the CF lung depends on the production of special chemicals that might be made only by very few types of bacteria. If that is true, medicines that interfere with those chemicals could treat the lung infections that cause trouble for nearly all people with CF. The investigators wish to study the production of several potentially critical chemicals by the respiratory bacteria and to examine the effect of those chemicals on the makeup of the entire community of bacteria. To detect all the bacteria in that community, the investigators will use new methods that use bacterial genetic information and can detect hundreds of different types of bacteria in respiratory samples of individual CF patients.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Cystic Fibrosis
* 2 to 55 years of age

Exclusion Criteria:

* None

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cystic fibrosis patients will be contacted during clinical care visits and inpatient hospitalizations.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hosptital, Boston, Boston, Massachusetts, United States